CLINICAL TRIAL: NCT00634725
Title: Randomized Multicenter Phase III Study in Patients With Locally Advanced Adenocarcinoma of the Pancreas: Gemcitabine With or Without Chemoradiotherapy and With or Without Erlotinib. Intergroup Study
Brief Title: Gemcitabine With or Without Capecitabine and/or Radiation Therapy or Gemcitabine With or Without Erlotinib in Treating Patients With Locally Advanced Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000589283; GERCOR-LAP-07-D07-1; EU=20827; ROCHE-GERCOR-LAP-07-D07-1; EudraCT- 2007-001174-81
Record Dates: First submitted 2008-03-12; First posted 2008-03-13 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2012-11

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Erlotinib Hydrochloride; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (A1) - Gemcitabine (Active Comparator): Gemcitabine 2 months, then stop until progression
  Interventions: Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis
- Arm 2 (B1) Gemcitabine + Erlotinib (Experimental): B1 Gemcitabine + Erlotinib (100mg/d) 2 months, then erlotinib maintenance (150 mg/d)until progression
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis
- Arm 3 (A2) CRT (Experimental): A2 CRT then stop until progression
  Interventions: Drug: capecitabine; Other: laboratory biomarker analysis; Radiation: radiation therapy
- Arm 4 (B2) CRT then erlotinib (Experimental): B2 CRT then erlotinib maintenance (150mg/d) until progression
  Interventions: Drug: capecitabine; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis; Radiation: radiation therapy

INTERVENTIONS:
Drug: capecitabine
  Arms: Arm 3 (A2) CRT; Arm 4 (B2) CRT then erlotinib
Drug: erlotinib hydrochloride
  Arms: Arm 2 (B1) Gemcitabine + Erlotinib; Arm 4 (B2) CRT then erlotinib
Drug: gemcitabine hydrochloride
  Arms: Arm 1 (A1) - Gemcitabine; Arm 2 (B1) Gemcitabine + Erlotinib
Other: laboratory biomarker analysis
Radiation: radiation therapy
  Arms: Arm 3 (A2) CRT; Arm 4 (B2) CRT then erlotinib

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known which regimen of chemotherapy with or without erlotinib and/or radiation therapy is most effective in treating pancreatic cancer.

PURPOSE: This randomized phase III trial is studying giving gemcitabine together with or without capecitabine and/or radiation therapy to see how well it works compared with giving gemcitabine together with or without erlotinib in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether administrating chemoradiotherapy in patients whose tumor is controlled after 4 months of induction chemotherapy (CT) increases survival compared with continuation of the same CT in patients with unresectable, locally advanced adenocarcinoma of the pancreas.

Secondary

* To assess whether erlotinib hydrochloride combined with gemcitabine hydrochloride and administered as maintenance treatment increases progression-free survival compared with gemcitabine hydrochloride alone and without maintenance treatment.
* To evaluate the response rate in the CT and chemoradiotherapy (CRT) arms.
* To evaluate tolerance to erlotinib hydrochloride as maintenance treatment after the end of CT or CRT.
* To study the predictive molecular factors (i.e., survivin, K-ras, EGFR, PTEN, or AKT) of survival.

OUTLINE: This is a multicenter study. Patients in the first randomization are stratified according to center and ECOG performance status (0-1 vs 2). Patients in the second randomization are stratified according to center and initial treatment arm (I vs II).

* First randomization: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43. Following the first evaluation, patients continue to receive gemcitabine hydrochloride on days 57, 64, 71, 85, 92, and 99 for a total of 4 months.
  * Arm II: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43. Following the first evaluation, patients continue to receive gemcitabine hydrochloride on days 57, 64, 71, 85, 92, and 99. Patients also receive oral erlotinib hydrochloride once daily for 4 months.

After completion of treatment in the first randomization proceed to the second randomization.

* Second randomization: Patients are randomized to 1 of 4 treatment arms.

  * Arm I: Patients continue gemcitabine hydrochloride as in arm I in the first randomization on days 113, 120, and 127 and on days 141, 148, and 155 for 2 months in the absence of disease progression.
  * Arm II: Patients continue gemcitabine hydrochloride as in arm II in the first randomization on days 113, 120, and 127 and on days 141, 148, and 155 and oral erlotinib hydrochloride daily for 2 months followed by erlotinib hydrochloride alone as maintenance therapy in the absence of disease progression.
  * Arm III: Patients receive oral capecitabine twice daily and undergo radiotherapy beginning on day 127, 5 days a week, for 6 weeks, in the absence of disease progression.
  * Arm IV: Patients receive oral capecitabine twice daily and undergo radiotherapy beginning on day 127, 5 days a week, for 6 weeks. Beginning 15 days after completion of CRT, patients receive a reintroduction of oral erlotinib hydrochloride alone once daily in the absence of disease progression or unacceptable toxicity.

Tumor tissue will be analyzed for the relationship between biological markers and resistance to treatment.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas meeting the following criteria:

  * De novo locally advanced disease
  * Unresectable disease
  * Stage III according to the UICC classification

    * No distant metastases
    * No localized stage IA-IIB or metastatic stage IV disease according to UICC classification
  * Not considered for curative resection after pluridisciplinary discussion

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Polynuclear neutrophils ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)

  * For patients who have had a recent biliary drain and whose bilirubin is descending, a value of ≤ 3 times ULN is acceptable
* Creatinine ≤ 2 mg/dL
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* Albumin ≥ 25 g/L
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of therapy

Exclusion criteria:

* Diarrhea ≥ grade 2 and/or uncontrolled diarrhea
* Affiliated with a social security regime
* Unable to follow instructions for psychological, familial, or geographical reasons
* Allergic to one of the ingredients in erlotinib hydrochloride
* Cancer within the past 5 years, except for in situ cancer of the neck of the uterus or basal cell skin cancer
* Severe infection
* Ophthalmic disease (i.e., inflammation, keratopathy, or infection)
* Symptomatic coronary or cardiac insufficiency, myocardial infarction, or stroke within the last 6 months
* Unable to take oral treatments
* Gastrointestinal disorders that could be associated with absorption disorders
* Untreated gastric or duodenal ulcer

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy (including abdominal radiotherapy) or chemotherapy for any reason
* No prior anti-epidermal growth factor-receptor therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | from the date of the first randomization to the date of patient death,due to any cause, or to the last date the patient was known to be alive, assessed up to 8 years after the beginning of the study
  an interim analysis is planned when 196 deaths will be observed

SECONDARY OUTCOMES:
Progression-free survival | time from the date of the first randomization to the date of progressive disease or death, assessed up to 8 years after the beginning of the study.
Relationship between biological markers and survival | From baseline to death, assessed up to 8 years after the beginning of the study
  1 biopsy/patient of the pancreas before treatment
tolerance to erlotinib | from start of treatment until the event has resolved or stabilized or until death
  To evaluate tolerance to erlotinib as maintenance treatment after the end of CT or CRT.
  During each visit, any adverse events will be noted and graded according to version 3 of the NCI-CTCAE. Any adverse events that persist at the end of the CTI will be followed up until they disappear.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Hammel, MD, PhD, Principal Investigator — Hopital Beaujon
Locations (72):
- France (72):
  - Centre Radiotherapie Oncologie Moyenne Garonne, Agen
  - Centre Hospitalier d'Aix en Provence, Aix-en-Provence
  - Centre Paul Papin, Angers
  - Polyclinique Sainte Marguerite, Auxerre
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Hopital Duffaut, Avignon
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Centre Hospitalier de Beauvais, Beauvais
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital de Beziers, Béziers
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - CHU de Caen, Caen
  - Polyclinique Du Parc, Caen
  - Hopital Beaujon, Clichy
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Compiegne, Compiègne
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier de Dax, Dax
  - Centre Hospitalier de Digne les Bains, Digne-les-Bains
  - Hopital Du Bocage, Dijon
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Draguignan, Draguignan
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - Hopital Louis Pasteur - Le Coudray, Le Coudray
  - Centre Hospitalier Universitaire de Bicetre, Le Kremlin-Bicêtre
  - Clinique Victor Hugo, Le Mans
  - Hopital Robert Boulin, Libourne
  - Polyclinique Du Bois, Lille
  - Polyclinique des Quatre Pavillons, Lormont
  - Centre Hospitalier St. Joseph St. Luc, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Hopital de la Croix Rousse, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Centre Gray, Maubeuge
  - Centre Hospitalier Chanaux, Mâcon
  - Centre Hospitalier de Meaux, Meaux
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier de Montelimar, Montélimar
  - C.H.U. de Nimes - Groupe Hospitals-Universitaire Caremeau, Nîmes
  - Clinique De Valdegour, Nîmes
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Saint Joseph, Paris
  - Hopital Tenon, Paris
  - Centre Catalan d'Oncologie, Perpignan
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Hopital Rene Dubos, Pontoise
  - CHU - Robert Debre, Reims
  - Hopital Charles Nicolle, Rouen
  - Centre Hospitalier, Saint-Omer
  - Centre Hospitalier de Tarbes, Tarbes
  - Centre Hospitalier Regional Metz Thionville, Thionville
  - CHRU de Tours - Hopital Trousseau, Tours
  - Nouvelle Clinique Generale, Valence
  - Centre Hospitalier Bretagne Atlantique, Vannes

REFERENCES:
- [Derived] Hammel P, Huguet F, van Laethem JL, Goldstein D, Glimelius B, Artru P, Borbath I, Bouche O, Shannon J, Andre T, Mineur L, Chibaudel B, Bonnetain F, Louvet C; LAP07 Trial Group. Effect of Chemoradiotherapy vs Chemotherapy on Survival in Patients With Locally Advanced Pancreatic Cancer Controlled After 4 Months of Gemcitabine With or Without Erlotinib: The LAP07 Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1844-53. doi: 10.1001/jama.2016.4324. PMID 27139057